CLINICAL TRIAL: NCT02288221
Title: SafEE : Safe & Easy Environment at Home for Patients Presenting a Frail Syndrome
Brief Title: Safe & Easy Environment at Home for Patients Presenting a Frail Syndrome
Acronym: SafEE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 14-PP-04
Record Dates: First submitted 2014-08-19; First posted 2014-11-11 (Estimated); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Cognitive Deterioration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- With non pharmacological therapeutic (Experimental): Installation of ICT at patient's home
  Interventions: Other: Patient's answer with non pharmacological therapeutic
- Without non pharmacological therapeutic (Active Comparator): No change at patient's home
  Interventions: Other: Patient's answer without non pharmacological therapeutic

INTERVENTIONS:
Other: Patient's answer with non pharmacological therapeutic — Installation at patient's home of :
  * aromatherapy
  * music therapy
  * cognitive training in multimedia application offering cognitive games
  Arms: With non pharmacological therapeutic
Other: Patient's answer without non pharmacological therapeutic — No installation at patient's home
  Arms: Without non pharmacological therapeutic

SUMMARY:
All over the world the increasing prevalence of chronic disorders and its impact on functional decline is challenging the sustainability of health care systems. Older individuals also frequently experience the reversible "frailty syndrome", which overlaps with chronic diseases, increasing incidence of disability.

Building a global system aiming to take in charge all causes leading to loss of autonomy is a rather complicated task involving numerous Information and Communication technologies (ICT) solutions which are not always easy to use in everyday life.

The SafEE (Safe Easy Environment) project aim is to improve the safety, autonomy and quality of life of older people at risk.

The SafEE project develop non pharmacological therapeutic through diferent ICT (stimulation aromatherapy automatic fragrance, training interface based on Kinect sensor...) .

The goal of this study is to validate the acceptability, sensitivity and efficacy of the systems.

DETAILED DESCRIPTION:
The non pharmacological therapeutic will be install at patient's home :

* aromatherapy,
* music therapy,
* cognitive training in multimedia application offering cognitive games.

Also smart phone will be given to the patient :

* to help him move with a geolocation application,
* to remind him of his daily needs (shopping lists, people to call, etc ...) with an alert apllication.

ELIGIBILITY:
Inclusion Criteria:

* Male or female age ≥ 60 years with memory complaint
* Score at the Mini Mental Test (MMSE) ≥ 26.
* Score at the Clinical Dementia Rating Scale (CDR) ≤ 0.5.

Exclusion Criteria:

* Sensory defect (visual or olfactory) preventing the patient to perfectly meet therapeutic solutions.
* Prescription new psychotropic medication (hypnotic, anxiolytic, antidepressant, antipsychotic) in the week preceding the assessment.
* Subject epileptic.
* Subject vulnerable

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2015-06-04 (Actual); Primary Completion 2017-07-05 (Actual); Study Completion 2017-07-05 (Actual)

PRIMARY OUTCOMES:
Time spent by the patient using the non-therapeutic solutions | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Renaud DAVID, Dr, Study Director — Centre Hospitalier Universitaire de Nice
Locations (1):
- Institut Claude Pompidou, Nice, France